CLINICAL TRIAL: NCT02418975
Title: Pre-operative Very Low-calorie Protein-based Versus Hypocaloric Enteral Nutrition to Improve Intra- and Post-operative Outcomes of Severely Obese Patients Undergoing Bariatric Surgery
Brief Title: Pre-operative Very Low-calorie Protein-based Versus Hypocaloric Enteral Nutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Giuseppe Moscati Hospital (Other)
Responsible Party: Principal Investigator, Giuseppe Castaldo, Physician, San Giuseppe Moscati Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CECN/132
Record Dates: First submitted 2015-03-19; First posted 2015-04-17 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Perioperative/Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Very low-calorie protein-based diet (Experimental): Patients will receive a homemade very low-calorie (~5 kcal/kg of ideal body weight /day) protein-based formula (milk proteins; 1.2 g per kilogram of ideal body weight) for 4 weeks by a polyurethane nasogastric feeding tube.
  Interventions: Other: Very low-calorie protein-based diet
- Hypocaloric diet (Active Comparator): Patients will receive a commercial balanced enteral formula (~20 kcal/kg of ideal body weight /day; protein content, 1.0 g per kilogram of ideal body weight) for 4 weeks by a polyurethane nasogastric feeding tube.
  Interventions: Other: Hypocaloric diet

INTERVENTIONS:
Other: Very low-calorie protein-based diet — Patients will receive a homemade very low-calorie (~5 kcal/kg of ideal body weight /day) protein-based formula (milk proteins; 1.2 g per kilogram of ideal body weight) for 4 weeks by a polyurethane nasogastric feeding tube.
  Arms: Very low-calorie protein-based diet
Other: Hypocaloric diet — Patients will receive a commercial balanced enteral formula (~20 kcal/kg of ideal body weight /day; protein content, 1.0 g per kilogram of ideal body weight) for 4 weeks by a polyurethane nasogastric feeding tube.
  Arms: Hypocaloric diet

SUMMARY:
Pre-operative weight loss can reduce the risk intra- and post-operative complications but no optimal pre-operative weight loss strategy has been investigated. Very-low-calorie diets (VLCDs) were proven to results in higher metabolic improvements in the short-term than balanced, hypocaloric diets. Therefore, the aim of the study is to investigate whether a VLCD results in lower intra-and post-operative complications compared to a hypocaloric diet. However, to achieve a optimal compliance in patients having experienced multiple dietary intervention failures, administration of the intervention will be performed by the enteral route using a naso-gastric feeding tube.

DETAILED DESCRIPTION:
Bariatric surgery is an important treatment strategy for obese patients having failed multiple diet-induced weight loss attempts. On the other hand, severly obese patients have also a high risk of both intra- and post-operative complications. Pre-operative weight loss can reduce these risks but no optimal pre-operative weight loss strategy has been investigated. Very-low-calorie diets (VLCDs) were proven to results in higher metabolic improvements in the short-term than balanced, hypocaloric diets. Therefore, the aim of the study is to investigate whether a VLCD results in lower intra-and post-operative complications compared to a hypocaloric diet. However, to achieve a optimal compliance in patients having experienced multiple dietary intervention failures, administration of the intervention will be performed by the enteral route using a naso-gastric feeding tube.

ELIGIBILITY:
Inclusion Criteria:

* patient candidate to laparoscopic bariatric surgery (gastric bypass or sleeve gastrectomy) after multi-disciplinary pre-operative evaluation
* Availability to long-term post-operative follow-up
* Normal kidney function serum creatinine ≤ 1,2 mg/dL and glomerular filtration rate ≥ 90 mL/min
* Normal liver function (aspartate amino-transferase and/or alanine amino-transferase and/or gamma glutamyl transferase < 2 x N)
* written informed consent

Exclusion Criteria:

* age <18 or >60 anni
* serum creatinine >1,2 mg/dl
* liver failure (Child-Pugh ≥ A)
* insuline-dependent diabetes mellitus
* atrioventricular block with QT > 0,44 ms
* Cardiac arrythmias
* Moderate-severe cardiac failure
* Hypokaliemia
* Chronic diarrhoea or vomitus
* 12-month previous cardio-vascular disease
* pregnancy and/or lactation
* current/previous neoplastic disease
* psychiatric disorders
* know gastro-intestinal diseases
* other controindications to enteral nutrition
* moderate-severe hypo-albuminemia (<3.0 mg/dL)
* 6-month previous diet-induced weight loss
* intragastric balloon
* unavailability to planned measurements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Surgery duration | End of surgery, an expected average of 3.5 hours
  from skin incision to wound closure

SECONDARY OUTCOMES:
Composite intra-operative complications | End of surgery, an expected average of 3.5 hours
  Hemorrhage, organ perforation or laceration, conversion to open surgery, stapler dysfunction
Composite post-operative complications | 30 days
  Any-type hemorrhage, any-type infections, wound dehiscence, anastomotic leak, organ dysfunction
Intra-operative bleeding | End of surgery, an expected average of 3.5 hours
Difficult intubation | Before surgery
Time to remove surgical drain | Hospital stay, an avarage of 9 days
Total drain fluid production | Hospital stay, an avarage of 9 days
Change of multiple biochemical parameters | End of dietary intervention, 28 days
  blood lipids, variables of glucose metabolism and growth-hormone axis
Change of multiple anthropometric parameters | End of dietary intervention, 28 days
  body mass index, body weight, waist and hip circumferences
Change in liver fibrosis | End of dietary intervention, 28 days
Change in liver volume | End of dietary intervention, 28 days
Change in visceral fat | End of dietary intervention, 28 days
Change of multiple body composition parameters | End of dietary intervention, 28 days
Change in handgrip strength | End of dietary intervention, 28 days
Change of multiple cardiac morpho-functional parameters | End of dietary intervention, 28 days
Length of hospital stay | Hospital stay, an avarage of 9 days
Composite complications of enteral feeding | End of dietary intervention, 28 days
  tube dysfunction, nausea, vomiting, diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Castaldo, MD, Principal Investigator — A.O.R.N. "San Giuseppe Moscati"
Locations (1):
- A.O.R.N. "San Giuseppe Moscati", Avellino, Italy

REFERENCES:
- [Background] Monaco L, Monaco M, Di Tommaso L, Stassano P, Castaldo L, Castaldo G. Aortomesenteric fat thickness with ultrasound predicts metabolic diseases in obese patients. Am J Med Sci. 2014 Jan;347(1):8-13. doi: 10.1097/MAJ.0b013e318288f795. PMID 24366220
- [Background] Sukkar SG, Signori A, Borrini C, Barisione G, Ivaldi C, Romeo C, Gradaschi R, Machello N, Nanetti E, Vaccaro AL. Feasibility of protein-sparing modified fast by tube (ProMoFasT) in obesity treatment: a phase II pilot trial on clinical safety and efficacy (appetite control, body composition, muscular strength, metabolic pattern, pulmonary function test). Med J Nutrition Metab. 2013;6(2):165-176. doi: 10.1007/s12349-013-0126-2. Epub 2013 May 30. PMID 24027606